CLINICAL TRIAL: NCT03634800
Title: Radiotherapy With Immunotherapy for Systemic Effect in Myeloma (RISE-M)
Acronym: RISE-M
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patient accruals.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1612017831
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Nivolumab; Immunotherapy; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Patients with multiple myeloma will receive Nivolumab intravenously at 240 mg every two weeks. Infusions will be given over 60 minutes (not bolus or IV push). Patients will continue to receive infusions every two weeks until disease progression or dose limiting toxicity is reached. Patients will receive radiation for 5 consecutive days. A dose of 6 Gy x 5 days will be administered. Patients may receive radiotherapy to an additional site at 12 weeks if they have stable disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- nivolumab/radiotherapy (Experimental): All eligible patients will receive immunotherapy (Nivolumab) plus radiotherapy (6 Gy x 5 fractions) to a targetable lesion.
  * Nivolumab 240 mg IV starts with the first radiotherapy fraction 240 mg IV every 2 weeks from first radiotherapy fraction until disease prograssion or dose limiting toxicity is reached
  * Radiotherapy Dose of 6 Gy x 5 days will be given (patients will receive 1 fraction over 5 days for a total of 5 fractions) during the first week of starting Nivolumab
  Interventions: Drug: Nivolumab 240mg; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Nivolumab 240mg — Patients with multiple myeloma will receive Nivolumab intravenously at 240 mg every two weeks. Infusions will be given over 60 minutes (not bolus or IV push). Patients will continue to receive infusions every two weeks until disease progression or dose limiting toxicity is reached.
  Other Names: Immunotherapy
Radiation: Radiation therapy — Patients will receive radiation for 5 consecutive days. A dose of 6 Gy x 5 days will be administered. Patients may receive radiotherapy to an additional site at 12 weeks if they have stable disease.

SUMMARY:
Eligible patients have multiple myeloma with measurable disease in the blood and a targetable soft tissue or bony lesion with radiotherapy. All eligible patients will receive immunotherapy (Nivolumab) plus radiotherapy, 6 Gy x 5 fractions, to a targetable lesion. Immunotherapy treatment starts with the first radiotherapy fraction. Nivolumab will be given every 2 weeks. Patients will have specified laboratory values measured bi-monthly and evaluated for response at 12 weeks as defined by International Myeloma Working Group Criteria. Patients will continue to receive their respective immunotherapy until disease progression or dose limiting toxicity is reached.

DETAILED DESCRIPTION:
All eligible patients will receive immunotherapy (Nivolumab) plus radiotherapy, 6 Gy x 5 fractions, to a targetable lesion. Immunotherapy treatment starts with the first radiotherapy fraction. Nivolumab will be given every 2 weeks. Patients will have specified laboratory values measured bi-monthly and evaluated for response at 12 weeks as defined by International Myeloma Working Group Criteria. Patients will continue to receive their respective immunotherapy until disease progression or dose limiting toxicity is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is, in the investigator's opinion, willing and able to comply with the protocol requirements.
2. Subject has given voluntary written informed consent before performance of any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care.
3. Must have received 2 consecutive cycles of systemic myeloma therapy.
4. Documented refractory or relapsed and refractory (R/R) multiple myeloma

   1. patients had less than minimal response, or had achieved at least a minimal response to previous treatment, but progressed within 6 months
   2. patients must have failed, be intolerant or are ineligible to treatment with an IMiD, proteasome inhibitor and anti-CD38 agent
5. Targetable plasmacytoma, either intra-or extramedullary that is visualized on imaging (PET/CT or MRI) and is causing symptoms (eg. pain, neurological compromise) or potential to cause symptom as per clinician's judgement; and measurable disease at screening, defined as one or more of the following:

   1. Serum IgG, IgA, or IgM M-protein ≥ 0.5 g/dL
   2. Urine M-Protein ≥ 200 mg excreted in a 24-hour collection sample
   3. Involved serum free light chain (sFLC) > 100 mg/L provided the FLC ratio is abnormal
6. Males and Females at least 18 years or legal age of consent per local regulations.
7. Women of childbearing potential (WOCBP) must have two negative serum or urine pregnancy tests (minimum sensitivity 25 mIU/mL or equivalent units of HCG). One 10-14 days prior to start of the study drug and one within 24 hours prior to the start of study drug.
8. Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.
9. No condition which would cause unacceptable risk.

Exclusion Criteria:

1. Subjects with solitary bone or extramedullary plasmacytoma as the only evidence of plasm cell dyscrasia.
2. Subjects with monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), Waldenstrom's macroglobulinemia, or POEMS syndrome (plasma cell dyscrasia with poly neuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
3. Subjects with active plasma cell leukemia (defined as either 20% of peripheral blood white blood cell count comprised of plasma/CD138+ cells or an absolute plasma cell count of 2 x 109/L).
4. Subjects within 100 days of stem cell transplantation.
5. Subjects within 4 weeks of surgery, unless cleared by surgeon.
6. Women who are of childbearing potential not complying to the above described contraceptive measures or are breastfeeding, and sexually active fertile men whose partners are WOCBP if they are not complying to the above described contraceptive measures.
7. Any uncontrolled or severe cardiovascular or pulmonary disease determined by the investigator, including:

   1. NYHA functional classification III or IV, congestive heart failure, unstable or poorly controlled angina, uncontrolled hypertension, arrhythmia, or myocardial infarction in the past 12 months
   2. Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
8. Active infection or know HBV/HCV/HIV.
9. Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
10. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of initiation of study drug. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
11. Previous radiotherapy to the area of the target area.
12. Prior exposure to immunotherapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Rossi, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital; Himanshu Nagar, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened and enrolled at 1 site in the US: Weill Cornell Medicine (NY, NY).
Groups:
- Nivolumab/Radiotherapy: All eligible patients will receive immunotherapy (Nivolumab) plus radiotherapy (6 Gy x 5 fractions) to a targetable lesion.
  * Nivolumab 240 mg IV starts with the first radiotherapy fraction 240 mg IV every 2 weeks from first radiotherapy fraction until disease prograssion or dose limiting toxicity is reached
  * Radiotherapy Dose of 6 Gy x 5 days will be given (patients will receive 1 fraction over 5 days for a total of 5 fractions) during the first week of starting Nivolumab
  Nivolumab 240mg: Patients with multiple myeloma will receive Nivolumab intravenously at 240 mg every two weeks. Infusions will be given over 60 minutes (not bolus or IV push). Patients will continue to receive infusions every two weeks until disease progression or dose limiting toxicity is reached.
  Radiation therapy: Patients will receive radiation for 5 consecutive days. A dose of 6 Gy x 5 days will be administered. Patients may receive radiotherapy to an additional site at 12 weeks if they have stable disease.
Period: Overall Study
Arm/Group | Nivolumab/Radiotherapy
Started | 6
Completed | 0
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Disease Progression | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 6 patients enrolled but 1 patient withdrew consent prior to starting treatment. 5 patients that enrolled and started treatment will be a part of the analysis population.
Arm/Group | Nivolumab/Radiotherapy
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 59.4 [26 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: To Determine Overall Response at 12 Weeks Using International Myeloma Working Group (IMWG) Criteria in Patients Will be Measured
Description: The primary aim is to estimate the overall response at 12 weeks using IMWG criteria. Per IMWG response criteria, Complete Response (CR) is defined as negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow; Very Good Partial Response (VGPR) is defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or > 90% reduction in serum M-protein plus urine M-protein level < 100 mg/24 h; Partial Response (PR) is defined as > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to < 200 mg/24 h, No change/Stable disease is defined as not meeting criteria for CR, VGPR, PR, or progressive disease; Progressive disease (PD) is defined as an increase of > 25% from lowest response value; Relapse is define as development of new soft tissue plasmacytomas or Definite increase in the size of existing plasmacytomas or bone lesions.
Time Frame: 12 weeks
Population: Out of the 5 patients that started treatment, only 3 patient made it to 12 weeks of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab/Radiotherapy
Number analyzed (Participants) | 3
Participants
  CR (complete response) | 0
  VGPR (Very Good Partial Response) | 0
  PR (Partial Response) | 0
  No change/Stable disease | 1
  PD (Progressive disease) | 2
  Relapse | 0

2. Secondary Outcome: To Determine the Median Progression Free Survival (PFS) Will be Assessed in Patients Treated With Immunotherapy and Radiotherapy.
Description: Median progression free survival for patients treated with immunotherapy and radiotherapy will be assessed. Progression free survival (PFS) will be defined as the time from first treatment day until objective or symptomatic progression. PFS will be defined as the time from first treatment day until objective or symptomatic progression and PFS will be assessed by Kaplan-Meier survival analysis and 95% confidence interval.
Time Frame: through study completion
Population: 4 patient progressed while on study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nivolumab/Radiotherapy
Number analyzed (Participants) | 4
days | 33.75 [21 to 56]

3. Secondary Outcome: To Determine the Median Overall Survival for Patients Treated With Immunotherapy and Radiotherapy Will be Assessed.
Description: Median overall survival for patients treated with immunotherapy and radiotherapy will be assessed. overall survival will be defined as the time from first treatment day until death. Overall survival will be assessed by Kaplan-Meier survival analysis and 95% confidence interval.
Time Frame: through study completion
Population: All patients withdrew consent after progressing, so no follow up survival data was collected (with the exception of 1 patient who only allowed for survival follow up after being taken off study for progression).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab/Radiotherapy
Number analyzed (Participants) | 1
months | 17.96 [17.96 to 17.96]

ADVERSE EVENTS:
Time Frame: Adverse event data is collected from the date of consent until patients withdraw consent. Patients removed from the the study treatment due to disease progression or unacceptable toxicity will be followed until their adverse event returns to baseline values or until study completion, whichever occurs first, unless they withdraw consent.
Description: 1 subject withdrew consent before to starting treatment and no AEs were collected, so only 5 subjects were evaluated for AEs.
Arm/Group | Nivolumab/Radiotherapy
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab/Radiotherapy (N=5)
Platelet count decreased (Investigations) | 1 (1) — Grade 4 platelet count decreased
Anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 3 Anemia
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3 back pain
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab/Radiotherapy (N=5)
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 3 Nausea
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) — Grade 1 Peripheral motor neuropathy
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1 Arthralgia
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1 Back pain
Fatigue (General disorders) | 1 (1) — Grade 1 Fatigue
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1 Myalgia
Bloating (Gastrointestinal disorders) | 1 (1) — Grade 1 Bloating
bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) — Grade 1 and Grade 2 Bone Pain
Vomiting (Gastrointestinal disorders) | 1 (1) — Grade 3 Vomiting
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 1 Diarrhea
Creatinine increased (Investigations) | 1 (1) — Grade 1 Creatinine increased
Alkaline phosphatase increased (Investigations) | 1 (1) — Grade 3 Alkaline phosphatase increased
Colitis (Gastrointestinal disorders) | 1 (1) — Colitis - grade unknown
pelvic pain (Reproductive system and breast disorders) | 1 (1) — Grade 1 Pelvic pain
Alanine aminotransferase increased (Investigations) | 1 (1) — Grade 2 Alanine aminotransferase increased
Aspartate aminotransferase increased (Investigations) | 1 (1) — Grade 2 Aspartate aminotransferase increased
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) — Grade 4 Hyperuricemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT03634800/Prot_SAP_000.pdf